CLINICAL TRIAL: NCT02700191
Title: Cardiovascular Diagnosis Using µ-Cor - an Interventional Pilot Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of interest by Investigators
Sponsor: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PCL-72-030
Record Dates: First submitted 2016-03-02; First posted 2016-03-07 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): For subjects in the Control arm, the parameters measured by the (µ-Cor) µ-Cor system will not be analysed or made available to the investigator.
- uCor (Experimental): For subjects in the Interventional arm, all of the parameters measured by the (µ-Cor) µ-Cor system will be available to the investigator and will remain blinded to the subjects. The investigator will use µ-Cor information to aid in therapy adjustment decisions during the study period.
  Interventions: Device: uCor

INTERVENTIONS:
Device: uCor
  Arms: uCor

SUMMARY:
Subjects that are being treated at the Congestive Heart Failure clinic in Nazareth will be given the µ-Cor system to be added to their standard care, and randomized 1:1 to an interventional arm or a control arm.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 20-90 years old.
* New York Heart Association (NYHA) class III-IV heart failure
* Followed by the Congestive Heart Failure (CHF) clinic in Nazareth
* Left ventricular ejection fraction <35%
* Requiring treatment with >40mg/day of furosemide* orally or with repeated bolus or intravenous infusion of furosemide* (*or equivalent bumetanide or torasemide).

Exclusion Criteria:

* Pregnancy
* Subjects who have received a heart transplant.
* Subjects who are unable or unwilling to follow the study requirements.
* Patients with allergies or skin sensitivities to electrode hydrogel and/or acrylic based adhesive.
* Patients with skin breakdown in areas on the chest where device and electrode placement is required

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
composite of all-cause death or hospitalizations due to heart failure in the Interventional arm compared to the Control arm. | 30 days to 3 months

IPD SHARING:
Plan to Share IPD: No